CLINICAL TRIAL: NCT01573975
Title: Comparison Between Ten Days Sequential Treatment (With Metronidazole or Tetracycline) and Ten Days Standard Triple Therapy of Helicobacter Pylori
Brief Title: Comparison Between Ten Days Sequential Treatment and Traditional Three Combined Treatment of Helicobacter Pylori
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Ming-Cheh Chen, Principal Investigator, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB097-76
Record Dates: First submitted 2012-04-04; First posted 2012-04-10 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; antibiotic resistance; sequential therapy; Taiwan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Seq-Metronidazole (Experimental): 10-day sequential therapy with metronidazole
  Interventions: Drug: 5RA-5RCM
- Seq-Tetracycline (Experimental): 10-day sequential therapy with tetracycline.
  Interventions: Drug: 5RA-5RCT
- Control (Active Comparator): 10-day standard triple therapy.
  Interventions: Drug: 10RCA

INTERVENTIONS:
Drug: 5RA-5RCM — rabeprazole 20mg b.i.d + amoxicillin 1000mg b.i.d x 5 days + rabeprazole 20mg b.i.d + clarithromycin 500mg b.i.d + metronidazole 500mg b.i.d x last 5 days.
  Other Names: Pariet x 10 days; Hiconcil x 1st 5 days then; Klaricid x last 5 days +; Flagyl x last 5 days
  Arms: Seq-Metronidazole
Drug: 5RA-5RCT — rabeprazole 20mg b.i.d + amoxicillin 1000mg b.i.d x 5 days + rabeprazole 20mg b.i.d + clarithromycin 500mg b.i.d + tetracycline 1000mg b.i.d x last 5 days.
  Other Names: Pariet x 10 days; Hiconcil x 1st 5 days then; Klaricid x last 5 days +; Acromycin x last 5 days.
  Arms: Seq-Tetracycline
Drug: 10RCA — rabeprazole 20mg b.i.d + clarithromycin 500mg b.i.d + amoxicillin 1000mg b.i.d x 10 days.
  Other Names: Pariet x 10 days; Klaricid x 10 days; Hiconcil x 10 days.
  Arms: Control

SUMMARY:
The purpose of this study is to compare the eradication efficacy of 10-day triple therapy with 10-day sequential therapy with tetracycline or metronidazole.

DETAILED DESCRIPTION:
Background: Antimicrobial resistance has decreased eradication rates for Helicobacter pylori infection worldwide.

Objective: To determine whether sequential treatment eradicates H. pylori infection better than standard triple-drug therapy for adults with dyspepsia or peptic ulcers in Taiwanese people.

Design: Randomized, single-blind, prospective controlled trial. Setting: A large tertiary referral hospital in eastern Taiwan. Patients: 450 patients with dyspepsia or peptic ulcers and infected by H. pylori.

Measurements: 13C-urea breath test, upper endoscopy, histologic evaluation, rapid urease test, bacterial culture, assessment of antibiotic resistance and CYP2C19 genotype of host.

Intervention: 450 patients with H. pylori infection are randomly assigned to receive one of the following therapeutic schemes: group A (5RA5RCT): rabeprazole (20 mg bid) plus amoxicillin (1 g bid) for 5 days, followed by rabeprazole (20 mg bid) plus clarithromycin (500 mg bid) and tetracycline (1g bid) for a further 5 days; group B (5RA5RCM): rabeprazole (20 mg bid) plus amoxicillin (1 g bid) for 5 days, followed by rabeprazole (20 mg bid) plus clarithromycin (500 mg bid) and metronidazole (500mg bid) for a further 5 days; group C as control: rabeprazole (20 mg bid) plus amoxicillin (1 g bid) and clarithromycin (500 mg bid.) for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* patient proved with infection of H. pylori in gastric mucosa
* adult with signed inform consent

Exclusion Criteria:

* woman in breast feeding or pregnancy.
* allergy to drugs used in study.
* three months without use of any antibiotic agents.
* patients under 20 years old.

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2009-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Eradication rate | 4 weeks after complete use of drug for treatment
  A negative post-treatment 13C-urea breath test or CLO test result at more than 4 weeks after complete use of drug for treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Cheh CHEN, MD, Principal Investigator — Buddhist Tzu Chi General Hospital
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan, Taiwan

REFERENCES:
- [Background] Graham DY, Abudayyeh S, El-Zimaity HM, Hoffman J, Reddy R, Opekun AR. Sequential therapy using high-dose esomeprazole-amoxicillin followed by gatifloxacin for Helicobacter pylori infection. Aliment Pharmacol Ther. 2006 Sep 1;24(5):845-50. doi: 10.1111/j.1365-2036.2006.03072.x. PMID 16918889
- [Background] Jafri NS, Hornung CA, Howden CW. Meta-analysis: sequential therapy appears superior to standard therapy for Helicobacter pylori infection in patients naive to treatment. Ann Intern Med. 2008 Jun 17;148(12):923-31. doi: 10.7326/0003-4819-148-12-200806170-00226. Epub 2008 May 19. PMID 18490667
- [Background] Vaira D, Zullo A, Vakil N, Gatta L, Ricci C, Perna F, Hassan C, Bernabucci V, Tampieri A, Morini S. Sequential therapy versus standard triple-drug therapy for Helicobacter pylori eradication: a randomized trial. Ann Intern Med. 2007 Apr 17;146(8):556-63. doi: 10.7326/0003-4819-146-8-200704170-00006. PMID 17438314
- [Background] Choi WH, Park DI, Oh SJ, Baek YH, Hong CH, Hong EJ, Song MJ, Park SK, Park JH, Kim HJ, Cho YK, Sohn CI, Jeon WK, Kim BI. [Effectiveness of 10 day-sequential therapy for Helicobacter pylori eradication in Korea]. Korean J Gastroenterol. 2008 May;51(5):280-4. Korean. PMID 18516011